CLINICAL TRIAL: NCT00198796
Title: Dose-finding Study of WS6788A, DS37-4 and H10407 Enterotoxigenic E. Coli (ETEC) Challenge Strains That Express Colonization Factors CS17 and CFA/I
Brief Title: Dose-finding Study of WS6788A, DS37-4 and H10407 Enterotoxigenic Escherichia Coli (ETEC) Challenge Strains
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Naval Medical Research Center (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CIR #193; CHR (H.22.03.10.28.A2) (Other: JHSPH IRB)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: We will initially study the effects of a 1x109 dose of H10407 (in 5 subjects) and then proceed to the dose-finding portion of the trial to study the effects of low (5x108) or higher doses (5x109) of the CS17 expressing strains (total of 20 subjects)

ARMS (1):
- H10407 (Experimental): H10407
  Interventions: Biological: H10407

INTERVENTIONS:
Biological: H10407 — The primary objective of the proposed clinical investigation is to validate a dose for ETEC H10407 that will cause diarrhea in 50% or more of subjects without causing high output diarrhea
  Other Names: Experimental

SUMMARY:
Five subjects will be admitted to the General Clinical Research Center (GCRC). The next day they will eat a light breakfast, fast for 90 minutes, ingest ETEC strain H10407, and fast for 90 more minutes. After this challenge they will be monitored closely , and all stools will be collected, graded and weighed. On Day 5, or sooner if indicated, they will begin antibiotics to eradicate the challenge strain. They will be scheduled for discharge on Day 7 but may leave a few days earlier if early antibiotic treatment is given.

Hypothesis:

A challenge dose of 10(9) colony forming unit (CFU) of ETEC strain H10407, will cause diarrhea in at least 60% of subjects.

DETAILED DESCRIPTION:
The rationale for validation H10407 in the challenge study proposed at Johns Hopkins University is that this initial challenge study will support additional challenge studies planned for the future. In these future studies, a bovine milk immunoglobulin containing high levels of antibodies specific for colonization factor antigen (CFA/I) or CFA/I-derived colonization factor will be investigated as a potential oral prophylaxis to neutralize subsequent challenge against CFA/I-expressing H10407 in the clinical setting. The goal here is therefore to validate a challenge dose of 1x109 h10407 organisms in the hands of the Johns Hopkins investigative team and to then use this dose in the future prophylaxis/challenge studies. Challenge doses equal to or comparable to the 1x109 dose proposed for the Johns Hopkins University (JHU) study have been used in 6 of the 9 challenge studies that have been done with the H10407 strain. The subsequent challenge studies using H10407 will be registered as part of other protocols.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults age 18 to 45 years old who are willing to participate, complete training on ETEC and diarrhea and procedures of the protocol, pass the test documenting knowledge of the study, and give informed consent.

Exclusion Criteria:

1. age<18 or >45 years
2. Chronic illness, chemical dependency, or significant medical illness as determined by the investigator.
3. immunosuppressive condition or IgA (Immunoglobulin A) deficiency
4. HIV antibody positive
5. hepatitis B surface antigen positive
6. hepatitis C antibody positive
7. travel to ETEC endemic area within 2 years
8. vaccination or other exposure to ETEC, cholera, or heat labile toxin (LT) toxin within 3 years
9. pregnancy as defined by + serum or urine - human chorionic gonadotropin (HCG) on the day before immunization
10. inability to pass the written examination
11. use of antibiotic, H2 blocking agent or proton pump inhibitor within 7 days of challenge
12. regular use of laxatives antacids or other agents to lower stomach acidity
13. significant abnormality in screening lav hematology and chemistry tests as determined by the investigator.
14. significant abnormality on EKG for those 40 to 50 years old as determined by the investigator.
15. allergy to quinolones, penicillin's and Bactrim.
16. abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2007-02-22 (Actual); Study Completion 2007-05-30 (Actual)

PRIMARY OUTCOMES:
To validate a dose for ETEC H10407 that will cause diarrhea in 50% or more of subjects without causing high output diarrhea, as determined by stool output volumes or signs and symptoms associated with hypovolemia. | 6 months

SECONDARY OUTCOMES:
To measure mucosal and systemic immune response to the somatic and toxin antigens of the H10407 strain. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robin McKenzie, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- General Clinical Research Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No